CLINICAL TRIAL: NCT02599779
Title: A Phase II Proof of Principle Study of the Activity of Pembrolizumab (MK-3475) in Combination With SBRT in Primary Tyrosine Kinase Inhibitor (TKI) Refractory Metastatic Kidney Cancer (mRCC) Patients
Brief Title: A Proof of Principle Study of Pembrolizumab With SBRT in TKI mRCC Patients
Acronym: OZM-065
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-065
Record Dates: First submitted 2015-09-09; First posted 2015-11-09 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Stage IV Renal Cell Cancer AJCC V7
Keywords: Renal cell cancer; SBRT; Pembrolizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm A (Experimental): Arm-A: Pembrolizumab will be started and Stereotactic Body Radiation Therapy will be given at the time of progression on pembrolizumab and pembrolizumab will be continued.
  Pembrolizumab will continue until progression as per immune related response criteria (irRC).
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy
- Treatment arm B (Experimental): Arm B: Pembrolizumab will be started. Stereotactic Body Radiation Therapy will be given before the 2nd course of pembrolizumab and pembrolizumab will be continued.
  Pembrolizumab will continue until progression as per immune related response criteria (irRC).
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — 200mg given intravenously over 30 minutes day 1 of every 3 week cycle until progression as per immune related response criteria
  Other Names: Keytruda, MK-3475
Radiation: Stereotactic Body Radiation Therapy — Dose and duration dependent on body site. In Arm A: SBRT given at the time of progression on pembrolizumab. In Arm B: SBRT given before the 2nd course of pembrolizumab.
  Other Names: SBRT

SUMMARY:
This study is designed as a phase-II proof of concept trial to investigate if a treatment strategy where stereotactic body radiation therapy (SBRT) is given with pembrolizumab is sufficiently active to warrant further investigation in randomized phase II or III studies. Metastatic renal cell cancer (mRCC) patients with PD-1 expressing immune cells are more likely to have larger more aggressive tumours and reduced survival and renal tumours that express PD-L1 are more aggressive with poorer outcome. Blocking this receptor/ligand interaction with monoclonal antibodies can restore the activity of tumour specific T-cells within the tumour with durable responses documented in early clinical trials in several tumour types including renal cell carcinoma. The study drug pembrolizumab is designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. SBRT will be given to the 1-3 most clinically significant lesions at the time of progression on pembrolizumab or at the 2nd course of pembrolizumab treatment in an effort to improve the activity of pembrolizumab. A total of 35 patients refractory to the approved first line therapy with a targeted drug (Sunitinib or Pazopanib) or untreated RCC patients with sarcomatoid differentiation will be enrolled on study. This group of patient has a poor outcome on any other 2nd line therapy and urgently need novel therapy.

DETAILED DESCRIPTION:
A phase II proof of concept, multi-centre, safety and efficacy study with a biomarker component to investigate if a treatment strategy where stereotactic body radiation therapy (SBRT) is given with pembrolizumab is sufficiently active to warrant further investigation in randomized phase II or III studies. The study will run for approximately 3 years, including 2 year of recruitment and 1 year of follow up. There will be two study arms. Enrollment of 15 patients into arm A will occur before the start of enrollment of the next 20 patients on arm B.

In arm A, pembrolizumab will be started and SBRT will be given to the 1-3 most clinically significant lesions only at the time of progression on pembrolizumab. Pembrolizumab will be continued after progression to detect if the addition of SBRT leads to stability or response in progressing lesions. After SBRT, untreated measurable disease must remain to assess the activity of continued pembrolizumab. Pembrolizumab and SBRT will continue until progression as per immune related response criteria (irRC). This cohort of patients will allow us to more clearly understand if SBRT does play a part in improving progression free survival when given in combination with pembrolizumab.

In arm B, pembrolizumab will be started and SBRT given before the 2nd course of pembrolizumab to the 1-3 most clinically significant lesions. After SBRT, untreated measurable disease must remain to assess the activity of pembrolizumab. The value of a treatment strategy that combines pembrolizumab and SBRT up-front is evaluated in this arm. Giving SBRT early to the most clinically significant cancer lesions may give pembrolizumab more time to work and may improve response by generating neo-antigens.

Patients will remain on study until progression as per irRC, withdrawal of consent or if they meet any of the premature withdrawal/discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Patients with a histologic confirmation of renal cell carcinoma with a clear cell component where the best response to first line TKI therapy (sunitinib, pazopanib, axitinib etc) is progression, or untreated RCC patients with sarcomatoid differentiation.
4. Evidence of measurable metastatic kidney cancer according to RECIST 1.1 criteria. Patients should have an adequate number of non-irradiated metastatic sites in order to adequately assess the activity of the pembrolizumab therapy.
5. Karnofsky performance status of ≥80.
6. Favorable (0 risk factors), intermediate (1-2 risk factors) and poor risk (3-6 risk factors) patients by the Heng prognostic model are eligible based on the number of the following risk factors present.
7. Demonstrate adequate organ function, all screening labs should be performed within 10 working days of the first dose of trial treatment.
8. Male subjects should agree to use an adequate method of contraception starting with the first dose of trial treatment through 120 days after the last dose of trial treatment.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of trial treatment. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. One to three extra-cranial metastases eligible for SBRT.

Exclusion Criteria:

1. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
2. Has had a prior monoclonal antibody within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
3. Has more than one previous targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately in the opinion of the investigator from the toxicity and/or complications from the intervention prior to starting trial treatment.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
5. Has known brain metastases and/or carcinomatous meningitis. Exceptions include patients who have completed treatment for brain metastases at least 3 months prior to starting treatment with pembrolizumab and remained stable and no longer require steroids to control brain edema.
6. Diagnosis of ataxia telangiectasia or active collagen vascular disease.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease, a history of non-infectious pneumonitis that required steroids, or current pneumonitis.
9. Has a known active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12; Primary Completion 2021-08 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival, as per irRC, for pembrolizumab, given with SBRT in metastatic RCC patients where progression is the best response to their first line therapy with a TKI, and in untreated patients with sarcomatoid differentiation. | up to 36 months

SECONDARY OUTCOMES:
Overall survival | up to 36 months
Objective response rate by immune related response criteria (irRC), and RECIST 1.1 criteria | up to 36 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Bjarnason, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario